CLINICAL TRIAL: NCT06785168
Title: The Effects of Machined Based Resistance Training in Older Patients With Chronic Heart Failure With Sarcopenia
Brief Title: The Effect of Resistance Training on Sarcopenia in Older Heart Failure Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kieu Nguyen Dang Phuong (Other)
Responsible Party: Sponsor-Investigator, Kieu Nguyen Dang Phuong, PhD student, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24590-DHYD
Record Dates: First submitted 2024-12-31; First posted 2025-01-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Sarcopenia in Elderly; Chronic Heart Failure
Keywords: sarcopenia; chronic heart failure; machine-based resistance training; age over 60; outpatient
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (US) (No Intervention): The participants will receive HF treatment as prescribed by cardiologists based on clinical guidelines. If participants have any additional medical conditions, their existing medications or treatments should continue. The prescribed medications should remain the same throughout the trial, with dosage adjustments only made if adverse events occur. The participants are also asked to maintain their usual physical activity, exercise routines, and dietary habits, without making changes outside of the study intervention. Researchers will contact incorrectly by phone weekly.
- Machine-based Resistance Training Group (Other): The participants will receive HF treatment as prescribed by cardiologists. If participants have any additional medical conditions, their existing medications or treatments should continue. They are also asked to maintain their usual physical activity, exercise routines, and dietary habits, without making changes outside of the study intervention. And they will train 3 nonconsecutive days/week during 8 weeks as follows: leg press and calf raise by Proxomed Compass 540 (Germany); leg curl, chest press, push up, seated row by HUR
  Interventions: Other: Machine-based Resistance Training

INTERVENTIONS:
Other: Machine-based Resistance Training — The participants will receive HF treatment as prescribed by cardiologists. If participants have any additional medical conditions, their existing medications or treatments should continue. They are also asked to maintain their usual physical activity, exercise routines, and dietary habits, without making changes outside of the study intervention. At the beginning, patients participating in resistance training should complete a pretest of one-repetition maximum (1-RM) to assess muscle strength, which will be used by a professional physical therapist to develop an individualized prescription. The specific movements are as follows: (1) leg press and (2) calf raise by Proxomed Compass 540 (Germany); (3) leg curl, (4) chest press, (5) push up, (6) seated row by HUR machine (US). During the 8 weeks, subjects will train 3 non-consecutive days/week with intensity 30%1-RM to 60% 1-RM, 3 sets/one excercise with 8-12 repetitions.
  Other Names: M-RT; A
  Arms: Machine-based Resistance Training Group

SUMMARY:
The goal of study is to evaluate the effects of an eight-week machine-based resistance training program on managing sarcopenia in older outpatients with chronic heart failure (HF) at Military Hospital 175.

DETAILED DESCRIPTION:
The participants will be randomly assigned to two groups: One group received machine-based resistance training (MRT) at the hospital, while the other group received usual care (US). The outcomes will be measured in the participants after 8 weeks including handgrip strength, gait speed, performance on the five-times sit-to-stand test.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 60 years old
* Meet the diagnostic criteria of 2019 AWGS2 sarcopenia, can be diagnosed once meeting (1) + (2) or (1) + (3) or (1) + (2) + (3): (1) Appendicular skeletal muscle mass (ASM): dual-energy X-ray absorptiometry (DXA) (male <7.0 kg/m², female <5.7 kg/m²). (2) Muscle strength: handgrip strength (male <28.0 kg, female <18.0 kg). (3) Physical performance: 6-meter walking speed <1.0 m/s.
* Meet the diagnostic criteria of heart failure following ESC 2021.
* Clearly understand the content and purpose of the study and sign the informed consent form.

Exclusion Criteria: There are contraindications for Exercise Testing in patients with stable heart failure according to ACSM 2022:

* Early stage after acute coronary syndrome (within the first 2 days)
* Unstable coronary artery disease
* Decompensated heart failure
* Acute venous thrombosis or recent arterial embolism (pulmonary or systemic)
* Acute myocarditis, pericarditis, endocarditis
* Aortic dissection of the valve
* Severe symptomatic aortic stenosis
* Acute systemic disease or fever
* Uncontrolled or life-threatening atrial or ventricular arrhythmias (including new-onset atrial fibrillation or flutter)
* Uncontrolled tachycardia (resting heart rate > 120 beats per minute)
* Third-degree AV block
* Uncontrolled diabetes
* Symptomatic orthostatic hypotension (> 20 mmHg)
* Gradually increasing fatigue during exercise or dyspnea at rest or with exertion within the past 3-5 days
* Significant myocardial ischemia at low workloads < 2 METs or 50W
* Relative contraindications according to ACSM 2022:
* Weight gain ≥ 1.8 kg in the past 1-3 days
* Simultaneous use of continuous or intermittent Dobutamine
* Decrease in blood pressure with exercise
* NYHA IV heart failure
* Complex ventricular arrhythmias at rest or with exertion
* Resting heart rate ≥ 100 bpm when lying down
* Comorbidities that limit exercise
* Severe obstructive hypertrophic cardiomyopathy
* Have participated in a cardiovascular rehabilitation program within the last 6 months
* Do not agree to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of muscle strength | Baseline and 8 weeks
  The change of muscle strength will be evaluated using handgrip strength, measured in kilograms. Each hand will be tested twice with a Jamar Hydraulic Hand Dynamometer (USA), and the highest value will be recorded.
The change of gait speed | Baseline and 8 weeks
  Gait speed is measured in meters per second. Participants will walk at their usual pace over a 6-meter distance, and gait speed will be calculated using the formula v = s/t, where t is the time in seconds and s is the distance (6 meters).
The change of the five-times sit-to-stand test | Baseline and 8 weeks
  The five-times sit-to-stand test is timed in seconds. Participants will sit in a chair without armrests, ensuring their back and lower legs are straight, with their arms crossed over their chest. They will then stand up and sit down as quickly as possible. The time is recorded using a stopwatch, beginning when the participants stand for the first time and ending when they sit down for the fifth time.

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Dang P Kieu, M.D., Study Chair — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (2):
- Vietnam (2):
  - Military Hospital 175, Ho Chi Minh City
  - University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No
Information Security